CLINICAL TRIAL: NCT03293901
Title: Skeletal Hormone and Calcium Kinetic Responses to Load Carriage Exercise in Females
Brief Title: Calcium Kinetic Responses to Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17-13-HC
Record Dates: First submitted 2017-08-10; First posted 2017-09-26 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Nutritional Status; Bones
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rest (No Intervention)
- Exercise (Active Comparator): Militarily relevant exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Treadmill exercise for 60 minutes with load carriage (weighted vest, 30% body weight) completed three times during the 6 day kinetic period.
  Arms: Exercise

SUMMARY:
This randomized cross-over study will identify physiological factors that underlie changes in bone metabolism that could affect skeletal injury risk, to include increases in parathyroid hormone (PTH) in response to militarily relevant exercise in females. The primary objective is to determine the hormone and calcium (Ca) response to multiple bouts of load carriage exercise in females. The investigators hypothesize that PTH will increase after multiple bouts of load carriage exercise and this increase will be due to disruption in Ca kinetics, specifically either a decrease in fractional intestinal Ca absorption (FCA) or changes in bone formation and/or resorption.

DETAILED DESCRIPTION:
Initial military training (IMT) results in increased risk of stress fracture, particularly for females as up to 21% of females may sustain a stress fracture during IMT, an incidence that is approximately 4-fold higher than that for males. Young female adults will undergo two separate study periods in random order, one will include exercise and the other will not. Each study period will use dual stable Ca isotope methodology in order to determine Ca kinetic responses to a militarily relevant exercise, and dietary intake will be controlled. Kinetic analyses will include fractional intestinal Ca absorption (FCA), Ca flux into bone (Vo+) and out of bone (Vo-), as well as renal Ca handling. Serial blood samples collected during the study periods will also be used to determine hormonal responses to exercise. The treadmill exercise will consist of a 60 minute timed trial with load carriage (30% body weight) completed three times during the 6 day kinetic period. At the start of the study, blood will be collected for analysis of Ca and bone-related genetic markers, and habitual food intake and exercise will be assessed. The information gathered from this trial will be used to identify physiological responses that can be targeted by future interventions designed to improve bone responses to training and decrease injury risk in female Warriors.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-42 years
* No current or prior military service
* Exercise 2-5 x/wk
* Stable body weight for 2 months (±5 lbs)
* Body mass index (BMI) between 19-26 kg/m2
* VO2max between 35-50 ml·kg-1·min-1
* Willing to discontinue use of dietary supplements and abstain from alcohol for the duration of the study
* Have not donated blood within the last 8 weeks

Exclusion Criteria:

* History of endocrine disorders (e.g., diabetes, uncontrolled thyroid dysfunction, hypoparathyroidism, or hyperparathyroidism)
* History of bone-modifying disorders (e.g., osteogenesis imperfecta, osteopetrosis, or rickets)
* History of cardiovascular or renal disease
* Pregnancy or lactation in the last 6 months
* Routine use of medications known to affect bone or calcium metabolism (e.g., thiazide diuretics, bisphosphonates, oral steroids)
* A very restrictive diet or severe food allergies

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility based on female anatomical sex characteristics
Enrollment: 21 (Actual)
Dates: Start 2018-06-16 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Hormone response and calcium kinetics | Exercise or rest will occur on days 0, 2, and 4 and measures will be taken daily days 0-4. After a washout period, measures will be repeated 1-4 weeks later on days 0, 2, and 4 with whichever intervention was not performed during the first study period.
  After dosing with dual stable calcium isotopes, changes in calcium kinetics (isotopic rations) will be measured in response to multiple bouts of a militarily relevant load carriage exercise or no exercise (rest) in females.

SECONDARY OUTCOMES:
Fractional calcium absorption | Bone measurement will be taken at baseline and FCA will be measured once during each intervention (exercise or rest) on day 0.
  Determine whether fractional Ca absorption (FCA) is associated with bone microarchitecture and strength in females undergoing multiple bouts of a militarily relevant load carriage exercise
Single nucleotide polymorphisms | SNP measurement will be taken at baseline and calcium measurements will be taken daily on days 0-4 when undergoing exercise and daily on days 0-4 when there is no exercise (rest).
  Evaluate whether single nucleotide polymorphisms (SNPs) previously identified to be associated with circulating 25OHD concentrations explain some of the variability in calcium kinetic responses to load carriage exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Gaffney-Stomberg, PhD, RD, Principal Investigator — United States Research Institute of Environmental Medicine
Locations (1):
- United States Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States